CLINICAL TRIAL: NCT00468455
Title: Postoperative Quality of Life: Development and Assessment of a Novel Tool to Assess Quality of Life Following Colorectal Surgery
Brief Title: Post-Op Quality of Life After Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Conor Delaney, MD, PhD, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: 10-05-17
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Colorectal Neoplasms; Colitis, Ulcerative; Diverticulitis; Colonic Polyps; Crohn Disease
Keywords: Colorectal Surgery; Abdominal Surgery; Diverticulitis; Colon Cancer; Rectal Cancer; Colon Polyp; Rectal Polyp; Crohn's Disease
MeSH Terms: conditions — Colorectal Neoplasms; Colitis, Ulcerative; Diverticulitis; Colonic Polyps; Crohn Disease; Colonic Neoplasms; Rectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Laparoscopic or open colorectal surgery — Application of a post-operative diary to be completed by subjects. The intervention is standard of care laparoscopic or open surgery.

SUMMARY:
The purpose of this study is to produce a user-friendly tool- in the form of a questionnaire - to accurately assess early quality of life in patients after abdominal colorectal surgery from the first day after surgery to 6 months after. The study will also compare this questionnaire to the other currently available assessment tools. Patients are invited to participate if they are undergoing abdominal colorectal surgery at University Hospitals of Cleveland.

DETAILED DESCRIPTION:
The purpose of this study is to produce a user-friendly tool to accurately assess early quality of life in postoperative patients following abdominal colorectal surgery in the early postoperative period (from surgery to 6 months) that is practical for routine application. The study will also compare this tool to the current available tools, namely the Short Form (SF-36), the short form inflammatory bowel disease questionnaire (IBDQ), the Cleveland Clinic Global Quality of Life (CGQOL). Patients will be invited to participate if they are undergoing abdominal colorectal surgery at University Hospitals of Cleveland.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years of age and older
* Subjects of either sex
* Subjects who will undergo any colorectal abdominal surgery at University Hospitals of Cleveland
* Subjects who agree to participate in the study program and provide written informed consent
* Diagnoses of Crohn's disease, ulcerative colitis, rectal or colon cancer, colon or rectal polyps and diverticulitis

Exclusion Criteria:

* Patients in the middle of three part surgery or had recent surgery (i.e., back for stoma closure for J-pouch)
* Patients with diagnosis of rectal prolapse, condyloma or any other condition that cannot be performed abdominally with an open or laparoscopic procedure
* Patient who have undergone major surgery within the month prior to this colorectal surgery
* Pregnant women, minors, psychiatric patients and prisoners

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo laparscopic or open procedures from the Deopartment of Surgery at University Hospitals of Cleveland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. | 1 month to 1 hour prior to surgery
  The aim of this study is to evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. We would like to use this survey to elucidate how quality of life of the patient is changed with the presence of an abdominal wall hernia.
Evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. | 2 weeks post operatively
  The aim of this study is to evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. We would like to use this survey to elucidate how quality of life of the patient is changed with the presence of an abdominal wall hernia.
Evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. | 4 weeks post operatively
  The aim of this study is to evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. We would like to use this survey to elucidate how quality of life of the patient is changed with the presence of an abdominal wall hernia.
Evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. | 6 months post-operatively
  The aim of this study is to evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. We would like to use this survey to elucidate how quality of life of the patient is changed with the presence of an abdominal wall hernia.
Evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients | 1 year post-operatively
  The aim of this study is to evaluate the quality of life in patients with abdominal wall hernias using a user-friendly survey that is designed specifically for this population of patients. We would like to use this survey to elucidate how quality of life of the patient is changed with the presence of an abdominal wall hernia.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Delaney, MD, PhD, Principal Investigator — University Hospitals of Cleveland/ Institute for Surgical Innovation
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States